CLINICAL TRIAL: NCT03945786
Title: Diagnostic Performance of Simultaneous Hybrid (18)F-fluoro-D-glucose (FDG) Positron Emission Tomography/Magnetic Resonance Imaging (PET/MRI) in the Preoperative Staging of Endometrial Carcinoma
Brief Title: Diagnostic Performance of Hybrid PET/MRI in the Staging of Endometrial Carcinoma
Status: Suspended | Type: Observational
Why Stopped: Recuriting inclusion and exclusion criteria will be changed as COVID-19.
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Wang Shijun, Director of Obstetrics and Gynecology Department, Xuanwu Hospital, Beijing
Other Study IDs: 首发2018-2-2013
Record Dates: First submitted 2019-05-09; First posted 2019-05-10 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Endometrial Carcinoma
Keywords: Hybrid PET/MRI
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Endometrial carcinoma (EC) is one of the most common gynecologic malignancy in China. EC is staged surgically according to the International Federation of Gynecology and Obstetrics (FIGO) system, including depth of myometrial invasion, cervical invasion, and the presence of lymph node metastases. The benefit of lymph node resection on the prognosis of low-risk EC patients is not definite. An accurate staging method preoperative is needed.The purpose of this study is to evaluate the effect of simultaneous hybrid PET/MRI in EC preoperative staging.

DETAILED DESCRIPTION:
The treatment of EC is mainly surgery, mostly comprehensive staging surgery (complete hysterectomy, bilateral adnexectomy, pelvic and para-aortic lymph node resection). Lymph node metastasis rate in the early low-risk EC patients (histologically graded G1 and G2, myometrium invasion depth <50%, primary tumor diameter <2 cm) is low (<4%). Lymph node resection has no clear benefit on the prognosis of low-risk EC patients, but will bring greater trauma to the patients.

Accurate preoperative assessment of EC staging plays a decisive role in the individualized surgical range for EC patients. Preoperative imaging can assist in optimal treatment planning. Through ultrasound, MRI, PET we always cannot accurately measure the depth of muscle infiltration, lymph node metastasis and extra-uterine lesions. The simultaneous hybrid PET/MRI technology combines the characteristics of MRI in high-resolution imaging of soft tissue and the advantages of PET in strong ability to identify tumor metastases, so it may be capable for more accurate staging.

ELIGIBILITY:
Inclusion Criteria:

* EC suspicious patients consent to diagnostic curettage
* Patients who pass standard clinical PET/MRI screening procedures
* Undergoing surgical staging and/or debulking at Xuanwu Hospital, Beijing

Exclusion Criteria:

* Allergy to (18)F-fluoro-D-glucose
* Contraindication to MRI scanning
* Pregnant or breast feeding patients
* Participation in any other clinical trial which may interfere with this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with irregular vaginal bleeding, abnormal vaginal discharge and/or other risk factors for EC undergoing diagnostic curettage.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-06-03 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value in the depth of endometrial infiltration | one month
  In EC identified cases, sensitivity, specificity, accuracy, and positive and negative predictive values will be calculated for depth of endometrial infiltration measured by regular staging method and hybrid PET/MRI method, adopting D&C pathological results as the gold standard.
Diagnostic value of the lymph nodes metastasis | one month
  In EC identified cases, sensitivity, specificity, accuracy, and positive and negative predictive values will be calculated for lymph nodes metastasis detected by regular staging method and hybrid PET/MRI method, adopting D&C pathological results as the gold standard.
Diagnostic value of the distant metastasis | one month
  In EC identified cases, sensitivity, specificity, accuracy, and positive and negative predictive values will be calculated for distant metastasis detected by regular staging method and hybrid PET/MRI method, adopting D&C pathological results as the gold standard.

SECONDARY OUTCOMES:
Detection of endometrial carcinoma by hybrid PET/MRI | one month
  In EC suspicious cases, sensitivity, specificity, accuracy, and positive and negative predictive values of hybrid PET/MRI for EC will be calculated, adopting D&C pathological results as the gold standard.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Stecco A, Buemi F, Cassara A, Matheoud R, Sacchetti GM, Arnulfo A, Brambilla M, Carriero A. Comparison of retrospective PET and MRI-DWI (PET/MRI-DWI) image fusion with PET/CT and MRI-DWI in detection of cervical and endometrial cancer lymph node metastases. Radiol Med. 2016 Jul;121(7):537-45. doi: 10.1007/s11547-016-0626-5. Epub 2016 Mar 31. PMID 27033474
- [Background] Kitajima K, Suenaga Y, Ueno Y, Kanda T, Maeda T, Takahashi S, Ebina Y, Miyahara Y, Yamada H, Sugimura K. Value of fusion of PET and MRI for staging of endometrial cancer: comparison with (1)(8)F-FDG contrast-enhanced PET/CT and dynamic contrast-enhanced pelvic MRI. Eur J Radiol. 2013 Oct;82(10):1672-6. doi: 10.1016/j.ejrad.2013.05.005. Epub 2013 May 30. PMID 23727380
- [Background] Nakajo K, Tatsumi M, Inoue A, Isohashi K, Higuchi I, Kato H, Imaizumi M, Enomoto T, Shimosegawa E, Kimura T, Hatazawa J. Diagnostic performance of fluorodeoxyglucose positron emission tomography/magnetic resonance imaging fusion images of gynecological malignant tumors: comparison with positron emission tomography/computed tomography. Jpn J Radiol. 2010 Feb;28(2):95-100. doi: 10.1007/s11604-009-0387-3. Epub 2010 Feb 26. PMID 20182843
- [Background] Li X, Zheng S, Chen S, Qin F, Lau S, Chen Q. Trends in gynaecological cancers in the largest obstetrics and gynaecology hospital in China from 2003 to 2013. Tumour Biol. 2015 Jul;36(7):4961-6. doi: 10.1007/s13277-015-3143-6. Epub 2015 Feb 4. PMID 25649977